CLINICAL TRIAL: NCT01721252
Title: Prospective Evaluation of a Proteomic Signature Developed to Identify Patients Likely to Benefit From Erlotinib (TarcevaTM), an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Used in the Treatment of Non-small Cell Lung Cancer
Brief Title: Tarceva. ICORG 08-41
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 08-41
Record Dates: First submitted 2012-10-24; First posted 2012-11-05 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; Erlotinib; TarcevaTM; proteomic signature
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aim of this study is to determine prospectively the value of a recently identified proteomic signature in identifying those patients with lung cancer, who are likely to benefit from and respond favourably to erlotinib therapy.

This is a prospective study of serum proteomics as a predictor of response to erlotinib therapy.

DETAILED DESCRIPTION:
Screening/Baseline

1. Routine blood tests (Haematology and Biochemistry) as per hospital practice
2. Research serum sample for proteomic studies (10ml blood sample)
3. Routine pre-treatment CT but with formal RECIST/WHO measurements of tumour size

2 months Post Commencement of Treatment with erlotinib: Routine CT with RECIST/WHO assessment

4 months Post Commencement of Treatment with erlotinib: Routine CT with RECIST/WHO assessment

1 year Post Commencement of Treatment with erlotinib (as per current standard of care): Routine CT with RECIST/WHO assessment

Response Assessment: CT scans at baseline, at 2 and 4 months post commencement of therapy and one year after treatment with erlotinib will be analyzed with the emphasis on identification of disease progression.

Follow Up: Subsequent follow-up as per routine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Any patient who is suited to receive CT scans as part of his/her routine care
* Ability to understand and the willingness to sign a written informed consent, given according to ICH/GCP, and national/local regulations. A signed informed consent must be obtained prior to any study specific procedures
* Planned treatment with erlotinib.

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients not foreseen to receive TarcevaTM treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient (18 years of age or older) diagnosed with non-small cell lung cancer at any stage who is to be treated with erlotinib.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-12; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Value of a recently identified proteomic algorithm | Change in CT scans taken at baseline, 2 and 4 months post commencement of therapy and one year after treatment with erlotinib will be analyzed with the emphasis on identification of disease progression.
  Routine CT with RECIST/WHO assessment

CONTACTS AND LOCATIONS:
Locations (7):
- Ireland (7):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St James Hospital, Dublin
  - The Adelaide & Meath Hospital, Dublin, Incorporating the National Children's Hospital, Dublin
  - Galway University Hospital, Galway
  - Mid-Western Regional Hospital, Limerick
  - Our Lady Of Lourdes Hospital, Drogheda, Louth